CLINICAL TRIAL: NCT06419049
Title: Impact of Standing Programs in Children With Spina Bifida: A Single Subject Design
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of St. Augustine for Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0819-275
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Spina Bifida
Keywords: Spina Bifida; Standing Device
MeSH Terms: conditions — Spinal Dysraphism

STUDY DESIGN:
Intervention Model Description: Single subject design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standing Program Intervention (Experimental): A single-subject study ABABA design will be used with dependent variables of passive range of motion, functional movement, functional skills performance, engagement, health related quality of life and gait velocity will be recorded repeatedly for the individual participants across time and with systematic manipulation of the independent variable, which is the standing home program intervention. The study will span 28 weeks for the intervention Stage 2, consisting of three baseline phases (A) of four weeks each and two home program intervention phases (B) of eight weeks each that alternate in an ABABA design.
  Interventions: Device: Altimate Medical EasyStand Bantam
- Reliability (No Intervention): Children will be assessed by two study investigators in two different sessions on the same day, with a washout period of 3 hours between sessions. Intrarater reliability will be determined by comparing rater's scores for each child. These sessions will include goniometric measurements of lower extremity passive range of motion and the 10-Meter Walk Test. Children will have the opportunity to rest or resume normal activities with a minimum of 3 hours between sessions. Interrater reliability will be determined based on the measurements in the same session by 2 different raters.

INTERVENTIONS:
Device: Altimate Medical EasyStand Bantam — Child will stand in stander 5 days per week for 60 min during each 8 wks intervention
  Arms: Standing Program Intervention

SUMMARY:
The purpose of this single-subject study is to investigate children with spinal bifida who have significant knee limitations in lower extremity passive range of motion to answer the following research questions:

1. Is a home standing program effective in reducing lower extremity passive range of motion limitations in children with Spina Bifida?
2. Does a home standing program change the quality of functional movement in children with spina bifida?
3. Does a home standing program change a child's performance in daily activities, mobility, and social/cognitive domains?
4. Does a home standing program change a child's health-related quality of life in children with spinal bifida?
5. Does a home standing program result in a change in gait velocity in children with Spina Bifida?

DETAILED DESCRIPTION:
Stage 1: Reliability Stage Each child will be assessed by two study investigators in two different sessions on the same day, with a washout period of 3 hours between sessions. Intrarater reliability will be determined by comparing rater's scores for each child. These sessions will include goniometric measurements of lower extremity PROM and the 10-Meter Walk Test. Children will have the opportunity to rest or resume normal activities with a minimum of 3 hours between sessions. Interrater reliability will be determined based on the measurements in the same session by 2 different raters.

Stage 2: Intervention Stage A single-subject study ABABA design will be used with dependent variables of passive range of motion, functional movement, functional skills performance, engagement, health-related quality of life and gait velocity will be recorded repeatedly for the individual participants across time and with systematic manipulation of the independent variable, which is the standing home program intervention. The study will span 28 weeks for the intervention Stage 2, consisting of three baseline phases (A) of four weeks each and two home program intervention phases (B) of eight weeks each that alternate in an ABABA design.

Regardless of the phase, the following primary measures will be assessed at baseline and every two weeks from the beginning until the conclusion of the study: Goniometric passive range of motion for all phases and hip and knee angle measures while standing in the stander during intervention phases and 10 meter walk test at preferred walking speed.

The following secondary measures will be assessed at baseline and every two weeks in phase A and every four weeks in phase B until the study's conclusion: Pediatric Neuromuscular Recovery Scale, Pediatric Evaluation of Disability Computer Adapted Test and Pediatric Quality of Life Inventory.

Nonintervention phase (A): The study investigator will meet face to face with the participant biweekly for 28 weeks to perform primary and secondary outcome measures. The Pediatric Neuromuscular Recovery Scale will be administered by the study investigator in person and scored by another investigator, who is an expert with the Pediatric Neuromuscular Recovery Scale, via video conference (not recorded).

Intervention phase (B): The study investigator will meet face to face with the participant biweekly for 28 weeks to perform outcome measures. The Pediatric Neuromuscular Recovery Scale will be administered by the study investigator in person and scored by another investigator via video conference. During the B phase, the study investigator will also provide parent instruction on the standing home program to ensure the parent and child can follow the home program. EasyStand will be providing the participants with the sit to stand stander for the duration of the intervention phases. A photo of the child in the stander will be taken by the investigator during each of these sessions and may be used in the dissemination of the project. The parent will keep a daily log of stander use and usual physical therapy-related activities. All of the measures will be analyzed to determine if there is a functional effect and if so, quantitative analysis methods will be used to determine the magnitude of the effect, and then the effect sizes will be combined to average intervention effects.

ELIGIBILITY:
Inclusion Criteria:

1) 5 to 12 years old, and 2) able to lay in a supine position on a plinth for testing and walk 10 meters. Participants will be excluded from the study if they have medical restrictions that contraindicate moving bilateral lower extremities through full passive range of motion (PROM), including but not limited to joint motion bony blocks, fractures before bone healing is complete, acute inflammatory or infectious process, disruption of soft tissue healing is likely, sharp, acute pain with joint movement or muscle elongation, hematoma or other soft tissue trauma, hypermobility and walking 10 meters.

Exclusion Criteria:

Participants will be excluded from the study if they have: 1) a diagnosis unrelated to MMC form of SB that limits standing, 2) a Modified Hoffer Scale level of 5, indicating an inability to ambulate. 3) medical restrictions that contraindicate standing, including but not limited to fractures and severe osteoporosis that precludes weight-bearing, and compromised cardiovascular or respiratory systems.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Goniometric Measurements | Assessed at baseline and every two weeks from the beginning until the conclusion of the study at 28 wks.
  A universal goniometer will be used to measure the child's hip and knee joint passive range of motion.
10 Meter Walk Test | Assessed at baseline and every two weeks from the beginning until the conclusion of the study at 28 wks.
  The 10MWTpref measures gait velocity in youth with neurological diagnoses while using an assistive device and wearing orthoses

SECONDARY OUTCOMES:
Pediatric Neuromuscular Recovery Scale (Peds NRS) | Assessed at baseline and every two weeks in the nonintervention phase and every four weeks in intervention phase until the study's conclusion at 28 wks.
  Assesses the quality of functional movement in children with spina bifida ages 1-12yrs. The Peds NRS examines the quality of sitting, upper extremity function, standing and walking
Pediatric Evaluation of Disability Computer Adapted Test (PEDI-CAT) | Assessed at baseline and every two weeks in the nonintervention phase and every four weeks in intervention phase until the study's conclusion at 28 wks
  Clinical assessment in children with spinal impairments that measures four domains: 1) Daily Activities, 2) Mobility, 3) Social/Cognitive, and 4) Responsibility to construct a description of a child's functional status in everyday life
Pediatric Quality of Life Inventory (PedsQL™) | Assessed at baseline and every two weeks in the nonintervention phase and every four weeks in intervention phase until the study's conclusion at 28 wks
  Measure of the HRQOL in children with chronic health conditions

CONTACTS AND LOCATIONS:
Locations (1):
- University of St. Augustine, San Diego, California, United States